CLINICAL TRIAL: NCT03080740
Title: The Efficacy and Safety Study of Clindamycin Palmitate Hydrochloride Dispersible Tablet for the Treatment of Bacterial Vaginosis
Brief Title: The Efficacy and Safety Study of Clindamycin Palmitate Hydrochloride Dispersible Tablet Treatment of Bacterial Vaginosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Yipinhong Pharmaceutical CO.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YPH-BV
Record Dates: First submitted 2017-03-06; First posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — clindamycin palmitate; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clindamycin palmitate hydrochloride (Active Comparator): Clindamycin palmitate hydrochloride dispersible tablet 300mg, oral after meal, twice daily, a total of 7days
  Interventions: Drug: Clindamycin palmitate hydrochloride dispersible tablet
- Metronidazole (Active Comparator): Metronidazole Tablet 400mg, oral after meal , twice daily, a total of 7days
  Interventions: Drug: Metronidazole Tablet

INTERVENTIONS:
Drug: Clindamycin palmitate hydrochloride dispersible tablet — 300mg, oral after meal, twice daily, a total of 7days
  Other Names: No other Names
  Arms: Clindamycin palmitate hydrochloride
Drug: Metronidazole Tablet — 400mg, oral after meal , twice daily, a total of 7days
  Other Names: No other Names
  Arms: Metronidazole

SUMMARY:
Randomized, double blind, positive drug parallel comparison, multi-centre clinical trial to assess the Efficacy and Safety of Clindamycin palmitate hydrochloride dispersible tablet for the treatment of bacterial vaginosis

DETAILED DESCRIPTION:
Treatment group: Clindamycin palmitate hydrochloride dispersible tablet . Control group: Metronidazole Tablet.

ELIGIBILITY:
Inclusion Criteria:

1. Patients clinically diagnosed with bacterial vaginosis, should meet the following criteria: vaginal Gram stain integration score (Nugent score) ≥7 points
2. Female patients aged 18 to 55 years old.
3. Patients signed the Informed Consent Form(ICF).

Exclusion Criteria:

1. Patients with vulvovaginitis caused by other infectional reasons such as vaginitis vulvovaginal candidiasis, trichomoniasis vaginitis.
2. Patients received systemic or vaginal antimicrobial therapy in a week before enrolled.
3. Patients with other vaginal or vulvar disorders which could effect the evaluation of efficacy.
4. Pregnant or lactating patients.
5. Menopausal women.

   Menopause definition: perimenopausal women stop menstruations for a year.
6. Women with diabetes.
7. Dependent on alcohol and could not prohibit during the study period.
8. Women with liver and kidney disfunction, blood disorders, mental illness or other serious diseases.
9. Women allergic to metronidazole, clindamycin.
10. With poor compliance.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Nugent score | From the first day of randomization to 4-10 and 23-33 days after the end,expected to be up to 33 days.Evaluate changes from baseline to the end of the study.
  score of Vaginal secretions for Gram stain

SECONDARY OUTCOMES:
The pH of vaginal secretions; | From the first day of randomization to 4-10 and 23-33 days after the end,expected to be up to 33 days.Evaluate changes from baseline to the end of the study.
  pH value
Leucorrhea routine examination | From the first day of randomization to 4-10 and 23-33 days after the end,expected to be up to 33 days.Evaluate changes from baseline to the end of the study.
  Vaginal cleanliness
Itching score | From the first day of randomization to 4-10 and 23-33 days after the end,expected to be up to 33 days.Evaluate changes from baseline to the end of the study.
  The severity of vulvar itching
Vaginal secretions | From the first day of randomization to 4-10 and 23-33 days after the end,expected to be up to 33 days.Evaluate changes from baseline to the end of the study.
  The amount of secretions

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Liu, MD, Study Chair — Peking University First Hospital; Shangrong Fan, MD, Principal Investigator — Peking University Shenzhen Hospital; Long Sui, MD, Principal Investigator — Affiliated Gynecology and Obstetrics Hospital of Fudan University; Ruifang An, MD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- Peking University first hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided